CLINICAL TRIAL: NCT07348562
Title: Omega-3 Fatty Acids, Inflammation and Attention Deficit Hyperactivity Disorder (ADHD) With AI (OmInADHDAI)- A Double-blind Randomized Controlled Trial of High Dose Omega-3 Fatty Acids in Children With ADHD With High Inflammation Status
Brief Title: Omega-3, Inflammation in ADHD With AI
Acronym: OmInADHDAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Pei-Chen Chang, Attending Physician, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH109-REC2-026
Record Dates: First submitted 2024-04-25; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Adhd
Keywords: children; inflammation; omega-3
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Inflammation | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: To investigate the effects of DHA, EPA and placebo in children and adolescents with ADHD
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Omega-3 (DHA) (Experimental): DHA supplementation
  Interventions: Dietary Supplement: Omega-3
- Omega-3 (EPA) (Experimental): EPA supplementation
  Interventions: Dietary Supplement: Omega-3
- Placebo (Placebo Comparator): olive oil
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 — Omega-3 PUFAs
  Arms: Omega-3 (DHA); Omega-3 (EPA)
Dietary Supplement: Placebo — Olive oil
  Arms: Placebo

SUMMARY:
This is a 12 week study to investigate the effects of omega-3 polyunsaturated fatty acids (PUFAs) in children with attention deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
This is a 12 week study to investigate the effects of omega-3 PUFAs in children (6-12 years-old) with ADHD.

The primary outcome will be the clinical symptoms The secondary outcomes will be inflammatory biomarkers, cognitive function and physiological markers such as heart-rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD (DSM-5) made by a child and adolescent psychiatrist.
* Age range: 6-12 years old at the time of enrollment.
* SNAP-IV (Mandarin Chinese Version):

Inattention subscale score > 12 or Hyperactivity/impulsivity subscale score > 12 or Total score > 24

* Drug-naïve or no ADHD medication use in the past 6 months.
* Signed informed consent required.

Exclusion Criteria:

* Intelligence quotient <80
* Comorbid other psychiatric disorders, such as autism spectrum disorder, anxiety disorder, conduct disorder, schizophrenia, mood disorder
* Comorbid physical disorders, such as thyroid dysfunction, cerebral palsy, coagulation disorders
* Currently using omega-3 supplements
* Allergy to omega-3

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Clinical Symptoms-Swanson, Nolan, and Pelham Rating Scale-4th Edition(SNAP-IV) | Baseline, week 1,2,4,8,12
  The SNAP-IV is used assess symptoms of ADHD (Attention Deficit Hyperactivity Disorder) in children and adolescents. It consists of a series of questions that rate the severity of behaviors such as inattention, hyperactivity, and impulsivity, based on teacher and parent observations. The scale includes both parent and teacher versions, allowing for a comprehensive view of a child's behavior in different environments. The scoring system rates each behavior on a 4-point scale from 0 (never or rarely) to 3 (very often), and higher total scores indicate more significant ADHD symptoms. The results help clinicians in diagnosing ADHD and monitoring treatment progress.

SECONDARY OUTCOMES:
Concentration of Peripheral Inflammatory Biomarkers | Baseline and week 12
  high-sensitivty C-reactive protein (hs-CRP) (milligram/Liter, mg/L) Interleukin (IL)-6 (picogram/milliliter, pg/mL)
Cognitive function-Continuous Performance Test (CPT) | Baseline and week 12
  CPT is used to assess attention and impulsivity in the subjects. It involves presenting a series of stimuli (usually letters or numbers) on a screen, where the participant must respond to certain targets and ignore others, assessing their ability to sustain attention over time and control impulses. The test helps identify attention deficits, impulsivity, and response inhibition, key areas impacted in ADHD.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Chen Chang, MD, PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University, Taichung, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No